CLINICAL TRIAL: NCT03539679
Title: TERVEYS JA LIIKUNTA PUOLUSTUSVOIMISSA
Brief Title: HEALTH AND EXERCISE IN THE DEFENSE FORCES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Jyvaskyla (Other); UKK Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R16189
Record Dates: First submitted 2018-04-25; First posted 2018-05-29 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Physical Condition, Minor Psychological Component
Keywords: Exercise, sickness absences, health, military fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention group and control group.
Who Masked: Participant
Masking Description: Exclusion criteria is that a volunteer must be health enough to have permission to take part in the military fitness tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encouraging physical activity (Experimental): Encouraging physical activity by using motion sensor and feedback.
  Interventions: Other: Encouraging physical activity.
- CONTROL GROUP (No Intervention): No intervention.

INTERVENTIONS:
Other: Encouraging physical activity. — Encouraging physical activity with motion sensor's feedback.
  Arms: Encouraging physical activity

SUMMARY:
The most important goal is to create a cost-effective, stimulating model for improving the employee's quality of life, work ability, and job satisfaction in the military operating environment. This is achieved by finding out how to activate an individual with the phone-based gaming and web-based feedback system to improve his physical condition. This study also tries to find out the adequate amount of physical activity to maintain the physical health of workers.

Personnel work ability, to work safe in service and effective operation capability of emergency forces require a worker's state of total well-being, in which the health and the physical condition are important parts. The changes in these affects the individual's fitness to military. This study develops a model to encourage an individual to carry out physical activity by himself. This will lead to reduce the sick leaves and improve the health and fitness.

Physical activity reduces morbidity. Professional soldiers must maintain their physical condition and skills. The study explores the optimum amount of working-age physical activity. It helps to maintain the working ability and one's fitness to field operations. With the help of the developed model it is possible cost-effectively activate a large number of employees to move more and to live more healthily.

DETAILED DESCRIPTION:
In this study it will be used motion sensors which are sending feedback to individuals mobile phone. Feedback is also given by email and in an interview after analyzing data from cloud service.

In the beginning of the study it will analyzed blood test, salivary test, body composition, height weight and basic motion. All volunteers are also answering a questionnaire.

There will be an intervention group and a control group. The intervention group will receive feedback during the all six months they are carrying the motion sensor.

After 6 and 12 months the basic analyzes will be repeated. Sick leaves and the changes in the muscular fitness test and changes in the 12-minutes running test will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Voluntaries armed forces workers.

Exclusion Criteria:

* Health enough to participate the military fitness test.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Better physical condition. | 6 months.
  12-minutes running test are measured.
Less sick leaves. | From past 12 months up to next 12 months.
  The amount of sick leaves are measured.

SECONDARY OUTCOMES:
Positive changes in the TELI v 1.0 questionnaire. | 6 months.
  Number of participants with better outcome in health habits (sleeping, eating, exercise).
Better physical condition. | 6 months.
  Muscular fitness test.

OTHER OUTCOMES:
Better physical condition. | 12 months.
  12-minutes running test are measured.
Better physical condition. | 12 months.
  Muscular fitness test.
Positive changes in the TELI v 1.0 questionnaire. | 12 months.
  Number of participants with better outcome in health habits (sleeping, eating, exercise).

CONTACTS AND LOCATIONS:
Overall Officials: KAI I PARKKOLA, PROF EMER, Study Director — PROF EMER, UNIVERSITY OF TAMPERE; HEIKKI KYRÖLÄINEN, PROF, Study Director — PROF, UNIVERSITY OF JYVÄSKYLÄ
Locations (1):
- Kai Parkkola, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No